CLINICAL TRIAL: NCT05760872
Title: Ffect of Acute Psychosocial Stress on Esophageal Sensitivity in Patients With Refractory Gastro-esophageal Reflux Disease and Healthy Volunteers
Brief Title: Effect of MIST on Esophageal Sensitivity: Pilot Study
Acronym: PilotMIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S65302-pilot
Record Dates: First submitted 2021-10-20; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Cortisol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Placement of an esophageal catheter: In this group we will assess the influence of placing an esophageal catheter on the cortisol levels in HV
  Interventions: Other: Placing esophageal probe

INTERVENTIONS:
Other: Placing esophageal probe — Placing an esophageal probe through the mouth

SUMMARY:
Influence of placing the esophageal probe on the cortisol response. Number of cortisol (non)responders and association of heart rate and subjective perception of stress with cortisol levels.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD), defined as the presence of symptoms or lesions that can be attributed to the reflux of gastric contents into the esophagus, is an increasingly prevalent condition in Western societies. The most typical symptoms are heartburn and regurgitation, however GERD can also manifest itself through a variety of other esophageal and extra-esophageal symptoms (e.g. chronic cough).

GERD patients can be divided into different categories based on upper endoscopy and pH or impedance-pH (MII-pH) monitoring. In the absence of lesions (esophagitis) during upper endoscopy, a pH or MII-pH monitoring will be performed. A first subcategory are patients with true GERD, characterized by an abnormal acid exposure and a positive or negative symptom association. The second and third category are patients with reflux hypersensitivity (RHS) and functional heartburn (FH)characterized by normal acid exposure on the MII-pH monitoring and a positive and negative symptom reflux association, respectively.

The basis for symptom generation/perception in GERD patients is not yet completely understood, but different mechanisms have been proposed including esophageal hypersensitivity, in which psychosocial stress is considered as a potential factor. This was shown in a study where 64% of the participants with heartburn reported that psychological factors, such as life stress, aggravate their symptoms (5). Furthermore, Fass et al. observed that auditory stress exacerbated symptom perception during esophageal acid perfusion. Moreover, our group investigated the effect of intravenous corticotrophin releasing hormone (CRH) on esophageal in healthy volunteers and showed that CRH is able to increase esophageal sensitivity to mechanical distention. Nevertheless, these previously performed studies in patients have some limitations: no measurable increase in cortisol (hypothalamo-pituitary-adrenal (HPA)-axis was not affected in these studies) and patients with RHS and FH - in whom the effect of stress is hypothesized to be the most relevant - were not included.

To induce moderate psychologic stress in the current study, the Montreal Imaging Stress Task (MIST) will be used. During this protocol, participants receive mental arithmetic challenges, together with social evaluative threat components from the program and/or the investigator (sham condition: threat components from the program and/or the investigator are absent). This MIST protocol can be used when investigating the effects of perceiving and processing psychosocial stress in the human brain in functional imaging studies.

Therefore, we want to investigate the relation between sensitivity to different stimuli (esophageal sensitivity) and psychosocial stress in healthy volunteers and patients (True GERD, RHS and FH).

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 to 65 years. All participants will receive and sign a copy of the informed consent before initiation of the study.

Exclusion Criteria:

* A history of any upper gastrointestinal (GI) symptoms, complaints or diseases;
* Prior history of esophageal or gastric surgery or endoscopic anti-reflux procedure;
* Psychiatric disorders;
* Concomitant use of other medication or treatments except for oral contraceptives;
* Use of medication altering GI motility;
* Pregnant or nursing women;
* History of drugs or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers with no or less experience with placing an esophageal probe
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
cortisol levels | every 15 minutes a saliva sample during 4.5 hours: at time points (in minutes) 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240, 255, 270
  Change in cortisol levels

SECONDARY OUTCOMES:
cortisol responders | up to 4 hours of cortisol measurement
  detect the number of cortisol responders

CONTACTS AND LOCATIONS:
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium